CLINICAL TRIAL: NCT00547859
Title: Correlation Between Microcirculatory Flow and Rectal Anaerobe Cellular CO2 Production in Patients After Cardiac Surgery
Brief Title: Relationship Between Microcirculatory Flow Alterations and Tissue Metabolism
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: EC Boerma, Medical Center Leeuwarden
Other Study IDs: TPO 503; ABR 19609
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Cardiac Surgery
Keywords: microcirculation; cardiac surgery; metabolism; capnometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to correlate microcirculatory flow and rectal anaerobe cellular CO2 production in patients after cardiac surgery. The hypothesis is that such a correlation exists.

DETAILED DESCRIPTION:
Sidestream Darkfield imaging is used to determine rectal microcirculatory flow in patients after postoperative cardiac surgery. At the same time PCO2 gap is established by monitoring rectal CO2 (tonometry) and arterial CO2 After initial enrollment and first analysis we also includes a control group with equal inclusion criteria for sublingual SDF imaging.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery
* informed consent
* age > 18

Exclusion Criteria:

* pregnancy
* off pump procedure
* rectal fecal contamination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post cardiac surgery patients in the first two hours of ICU treatment
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Relation between MFI (by SDF) and capno | 6 months

SECONDARY OUTCOMES:
Relevance of changes in flow and metabolism | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Department of ICU, Leeuwarden, PO Box 888, Netherlands

REFERENCES:
- [Background] Boerma EC, Mathura KR, van der Voort PH, Spronk PE, Ince C. Quantifying bedside-derived imaging of microcirculatory abnormalities in septic patients: a prospective validation study. Crit Care. 2005;9(6):R601-6. doi: 10.1186/cc3809. Epub 2005 Sep 22. PMID 16280059